CLINICAL TRIAL: NCT03227562
Title: Evaluation of Predictability of the Initial Response to a Low Dose of Risperidone on the Middle Term Efficiency in Anxious Subjects
Brief Title: Is Initial Response to Low Dose Risperidone Predictive for Outcome in Anxiety?
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: not enough patient
Sponsor: Marion Trousselard (Other Government)
Responsible Party: Sponsor-Investigator, Marion Trousselard, professor, Institut de Recherche Biomedicale des Armees
Organization: Institut de Recherche Biomedicale des Armees (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-000341-31
Record Dates: First submitted 2017-07-14; First posted 2017-07-24 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Anxiety State
Keywords: risperidone; anxiety; cognition; stress
MeSH Terms: conditions — Anxiety Disorders | interventions — Risperidone

STUDY DESIGN:
Intervention Model Description: All subjects are under 0.5mg risperidone (one group). Accordin to their response to treatment (responder vs. non responder) the 2 experimental groups will be created.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Responder (Other): The 2 arms will be created according to the early response to risperidone (responder vs. non responder)
  Interventions: Drug: RisperiDONE 0.5 MG
- Non responder (Other): The 2 arms will be created according to the early response to risperidone (responder vs. non responder)
  Interventions: Drug: RisperiDONE 0.5 MG

INTERVENTIONS:
Drug: RisperiDONE 0.5 MG — To be prescribed a 0.5mg risperidone treatment for anxiety is required to be enrolled.

SUMMARY:
Risperidone at low dosage is often used as treatment of acute anxiety symptom. However, patients may be either responder or not. Here we hypothesized that the early response to a low dose of risperidone is predictive to risperidone efficiency.

Subjects with acute anxiety symptoms (Hospital anxiety depression scale) and risperidone prescription would be proposed to be enrolled in the study. A check-up is made at D0, then the subjects begin the treatment (0.5mg risperidone). The same check-up is carried out on the following day (D1). The subjects fulfil a last check-up 12 week after the beginning of treatment (W12). During the D1-W12, the psychiatrist may changes the treatment.

DETAILED DESCRIPTION:
Risperidone at low dosage is often used as treatment of acute anxiety symptom. However, patients may be either responder or not. Here we hypothesized that the early response to a low dose of risperidone is predictive to risperidone efficiency.

Subjects with acute anxiety symptoms (Hospital anxiety depression scale) and risperidone prescription would be proposed to be enrolled in the study. After acceptation, the fulfil questionnaires (MINI, PCL-s-V) then they interacts with test on computers (PVT, 2nBack, Iowa gambling task) and give saliva and receive an actimetric watch (D0).

They begin the treatment on the evening (0.5mg risperidone/day). The following day, they come back to hospital and they fulfil the same tests, questionnaires and samples (D1).

12 week after, they come again to hospital to fulfil the same tests, questionnaires and samples (W12).

Between D1 and S12, the psychiatrist may change the treatment, adding other treatment or modifying risperidone treatment (increasing dosage up to 2mg/day or removing it).

ELIGIBILITY:
Inclusion Criteria:

* anxiety (score above 11 at anxiety scale of HADs)
* To have a prescription for 0.5 mg risperidone/day
* To give the consent
* To have a social protection
* To be adult (18-50 years)

Exclusion Criteria:

* Psychiatric antecedents
* any treatment for mental disease (antidepressant, anxiolytics, etc.)
* Ongoing neurological pathologies
* Scheduled surgery
* addiction
* pregancy
* known intolerance to risperidone
* participation to another biomedical study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Anxiety | changes between baseline and day 1 and between baseline and week 12
  score in Anxiety scale in the Hospital Anxiety Depression Scale (HADs)

SECONDARY OUTCOMES:
Type of anxiety | changes between baseline and day 1 and between baseline and week 12
  score in the Post-trauma CheckList 5

OTHER OUTCOMES:
Cognition | changes between baseline and day 1 and between baseline and week 12
  score in the Iowa Gambling Task

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand Lahutte, Principal Investigator — HIA Begin Paris
Locations (1):
- Marion Trousselard, Brétigny-sur-Orge, Not in US/Canada, France

IPD SHARING:
Plan to Share IPD: Undecided